CLINICAL TRIAL: NCT04943276
Title: A Novel Noninvasive Thermoregulatory Device for Postural Tachycardia
Brief Title: A Novel Noninvasive Thermoregulatory Device for Postural Tachycardia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Embr Labs, Inc. (Industry)
Responsible Party: Principal Investigator, Mitchell Miglis, Clinical Assistant Professor, Neurology and Neurological Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-59863
Record Dates: First submitted 2021-06-23; First posted 2021-06-29 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Postural Tachycardia Syndrome
Keywords: Thermoregulation
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Embr Watch (Experimental): Participants will receive the device and a technical onboarding video 3 days prior to study start to allow time for familiarization with the device and troubleshooting any technical questions or problems prior to study start. The study will consist of baseline measurements prior to using the Embr device and weekly outcome assessments at Week 1, 2, 3, and 4
  Interventions: Device: Embr Device

INTERVENTIONS:
Device: Embr Device — The Embr thermal device will be worn at all times from study start to the study endpoint.

SUMMARY:
The investigators hope to learn the feasibility and preliminary efficacy of the Embr device for improving thermal comfort in individuals with POTS and impaired thermoregulation. Feasibility will be assessed via usage of the Embr device and participant feedback. Preliminary efficacy measures will include temperature-related symptoms and temperature- related quality of life in individuals with POTS and impaired thermoregulation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POTS
* Participant self-report of heat or cold intolerance
* Willingness to wear the Embr device for 3 weeks, charging the device daily, and
* Have a working smartphone (iPhone 6 or greater; or Android 8.0 or greater
* Comfortable downloading and using the companion app on their phone
* Able to provide informed written consent
* Able to complete written questionnaires

Exclusion Criteria:

* Prior or current use of the study device
* Hypohidrosis, hyperhidrosis, or anhidrosis, as determined by sudomotor testing; peripheral neuropathy; perimenopausal, menopausal, postmenopausal state; temperature intolerance due to other medical disorders (i.e. malignancy, systemic autoimmune disease)
* Medications known to affect sweat function
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Compass-31 survey at study endpoint | Baseline and end of study ( 4 weeks)
  Compass 31 score ranges in value from 0 to 100. A score of 0 indicates no autonomic symptoms, while more-severe autonomic symptoms correspond to higher values.
Change from baseline in Pittsburg Sleep Quality Index (PSQI) at study endpoint | Baseline and end of study ( 4 weeks)
  PSQI score ranges in value from 0 to 21. A score of 0 indicates no sleep difficulties, while more-severe sleep difficulties correspond to higher values.
Change from baseline in Insomnia Severity Scale Index (ISI) at study endpoint | Baseline and end of study ( 4 weeks)
  Scale range is 0-28, with 0 indicating absence of insomnia and 28 indicating severe insomnia.
Temperature Quality of life Questionnaire | Week 1,2,3,4
Temperature related daily interference scale | Week 1,2,3,4
  Scale range is 0-100, with a higher score indicating more problems with thermoregulation.
OCEAN Temperature Related Psychogenic Questionnaire | Week 1,2,3,4

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Miglis, Principal Investigator — Stanford University
Locations (1):
- Stanford Neuroscience Health Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after de-identification. Only this de-identified data will be shared with the Embr team.
  PHI data will not be shared.
Time Frame: After study end. ( 1 Year after enrollment begins)
Access Criteria: Only Embr labs research team will have access to the de-identified data